CLINICAL TRIAL: NCT01458704
Title: Cancer Genome Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Cancer genome analysis
Record Dates: First submitted 2011-10-23; First posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Malignant Tumor
MeSH Terms: conditions — Neoplasms | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fresh frozen tumor tissue

GROUPS / COHORTS (1):
- fresh frozen tumor tissue: patients providing fresh frozen tumor tissue
  Interventions: Other: next generation sequencing

INTERVENTIONS:
Other: next generation sequencing — next generation sequencing (including targeted gene sequencing, exome sequencing, transcriptome sequenicing)

SUMMARY:
Next generation sequencing (including targeted gene seqeuncing, exome and transcriptome sequencing) will be performed from fresh frozen tumor samples to understand the genetic alteration of tumors and to aid in optimal selection of further therapeutic agents.

ELIGIBILITY:
Inclusion Criteria:

* patients with malignant tumor
* receiving or planning to receive chemotherapy
* with fresh frozen tumor tissue
* with informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with malignant tumor receiving or planning to receive chemotherapy with fresh frozen tumor tissue with informed consent
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
targeted sequencing of cancer-relate genes | 1 year
  Identification and characterization of genetic alteration in cancer tissue

CONTACTS AND LOCATIONS:
Overall Officials: Tae-You Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea